CLINICAL TRIAL: NCT00914459
Title: A Non-randomized, Open-label Study To Evaluate The Pharmacokinetics, Safety And Efficacy Of Refacto Af In Previously Treated Pediatric Subjects Less Than Twelve Years Of Age With Severe Hemophilia A (Fviii:c <1%).
Brief Title: Study Evaluating Safety And Efficacy Of Moroctocog Alfa (AF-CC) In Previously Treated Hemophilia A Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-4433; B1831005 (Other: Alias Study Number); 2008-008435-29 (EudraCT Number)
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Hemophilia A
Keywords: hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ; Factor VIII; Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moroctocog alfa (AF-CC) (Other): Open Label
  Interventions: Biological: Moroctocog alfa ( AF-CC); Procedure: Laboratory tests

INTERVENTIONS:
Biological: Moroctocog alfa ( AF-CC) — Dosing is at the discretion of the Investigator
  Other Names: ReFacto AF
Procedure: Laboratory tests — Factor VIII PK samples, Hematology, Chemistry and Coagulation testing, FactorVIII Inhibitor and Anti Factor VIII antibody

SUMMARY:
The study will be investigating pharmacokinetics, safety and efficacy in patients less than 12 years of age with severe hemophilia A that have been previously treated with Factor VIII products ( including blood products).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects less than 12 years of age with a documented history of severe hemophilia A (FVIII:C less than 1%).
* Subjects who are less than 6 years of age must have had at least 50 Exposure Days (EDs) to prior FVIII products (including blood products).
* Subjects who are equal to or greater than 6 years of age must have had greater than 150 EDs to prior FVIII products (including blood products).

Exclusion Criteria:

* For laboratory assessments, any measured Bethesda inhibitor titer equal to or greater than 0.6 BU, regardless of the laboratory normal range, or any Bethesda inhibitor titer greater than ULN for the testing laboratory at the time of screening.
* Any other bleeding disorder in addition to hemophilia A.
* Treatment with any investigational drug or device within 30 days before the time of signing the parental informed consent/assent form.
* Major surgery planned to occur during the course of the study.
* Regular (e.g., daily; every other day) use of agents or medications known to influence platelet function such as aspirin or certain nonsteroidal anti-inflammatory drugs (NSAIDS).
* Regular, concomitant therapy with immunomodulating drugs (e.g., intravenous immunoglobulin [IVIG], routine systemic corticosteroids), or currently receiving immune tolerance induction (ITI) for inhibitor treatment.
* The subject is receiving treatment for HIV or hepatitis infection (unless the subject is on a stable antiviral regimen [i.e., consistent treatment regimen for at least 3 months before the parental informed consent/assent form is signed]).
* Platelet count less than 100,000/µL.
* Prothrombin time (PT) equal to or greater than 1.25 x ULN, or international normalized ratio (INR) equal to or greater than 1.5.
* Known hypersensitivity to hamster protein.

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Kuopio University Hospital, Kuopio, Finland
- LTD Medinvesti- Institute of hematology and transfusiology, Tbilisi, Georgia
- Centro di Riferimento Regionale per la cura dell'Emofilia e delle Malattie Emorragiche Congenite, Parma, Italy
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Craiova, Craiova, Dolj
  - Sanador, Bucharest
- Serbia (2):
  - University Children's Hospital, Belgrade
  - Mother and Child Health Care Institute of Serbia "Dr Vukan Cupic", Belgrade
- Spain (4):
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Puerta del Mar, Cadiz, Spain
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza
  - Hospital La Paz, Madrid
- Karolinska Universitetssjukhuset-Solna, Stockholm, Sweden
- Turkey (Türkiye) (3):
  - Cukurova University Department of Pediatrics, Pediatric Hematology Division, Adana, Balcali/adana
  - Ege University Department of Pediatrics, Pediatric Hematology Division, Izmir, Bornova /izmir
  - Akdeniz Universitesi Tip Fakultesi, Antalya, Kampus
- Ukraine (2):
  - Komunalna ustanova "Zaporizka oblasna klinichna dytiacha likarnia", Zaporizhzhia, Ukraine
  - Derzhavna ustanova "Instytut patolohii krovi ta transfuziinoi medytsyny Natsionalnoi akademii medych, Lviv

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-4433&StudyName=Study%20Evaluating%20Safety%20And%20Efficacy%20Of%20Moroctocog%20Alfa%20%28AF-CC%29%20In%20Previously%20Treated%20Hemophilia%20A%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- ReFacto AF: Less Than 6 Years: Participants below 6 years of age were treated with IV injections of ReFacto AF at a dose and frequency prescribed by the investigator (minimum dose of 17 international units per kilogram [IU/kg] up to maximum dose of 51 IU/kg) as per local standard of care in accordance with the Summary of Product Characteristics (SmPC).
- ReFacto AF: 6 to Less Than 12 Years: Participants of 6 to 12 years of age were treated with IV injections of ReFacto AF at a dose and frequency prescribed by the investigator (minimum dose of 17 IU/kg up to maximum dose of 51 IU/kg) as per local standard of care in accordance with the SmPC.
Period: Overall Study
Arm/Group | ReFacto AF: Less Than 6 Years | ReFacto AF: 6 to Less Than 12 Years
Started | 18 | 19
Completed | 17 | 18
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Parent/Legal guardian request | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated analysis set included all enrolled participants who received at least 1 dose of ReFacto AF.
Groups:
- ReFacto AF: Less Than 6 Years: Participants below 6 years of age were treated with IV injections of ReFacto AF at a dose and frequency prescribed by the investigator (minimum dose of 17 IU/kg up to maximum dose of 51 IU/kg) as per local standard of care in accordance with the SmPC.
- Total: Total of all reporting groups
Arm/Group | ReFacto AF: Less Than 6 Years | ReFacto AF: 6 to Less Than 12 Years | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.6 (1.42) | 9.2 (1.47) | 6.5 (3.20)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Factor VIII Inhibitor Development
Description: Clinically significant factor VIII (FVIII) inhibitors were defined as a central laboratory confirmed positive inhibitor of greater than or equal to (>=) 0.6 Bethesda units (BU) using the Nijmegen modification of the Bethesda assay present at 2 consecutive blood draws within a 6-week interval and one of the following within 4 weeks before the initial or within 4 weeks following the second positive FVIII inhibitor sample collection: 1) the need for the participant to administer alternative hemostatic products in order to achieve sufficient efficacy, 2) >=2 events indicating a decrease in the efficacy of the study treatment. Percentage of participants who developed clinically significant Factor VIII inhibitor after study drug administration were reported.
Time Frame: Baseline up to Month 24
Population: Safety analysis population included all enrolled participants who received at least 1 dose of ReFacto AF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ReFacto AF: Less Than 6 Years | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 18 | 19
percentage of participants | 0.00 [0.00 to 18.53] | 0.00 [0.00 to 17.65]

2. Primary Outcome: Incremental Recovery
Description: Incremental recovery was the increase in circulating FVIII activity for every international unit (IU) of ReFacto AF administered per kilogram of body weight. It was measured in international units per deciliter (IU/dL) per international units per kilogram (IU/kg).
Time Frame: Days 1, 15, 50, Months 6, 18 and Final visit (up to Month 24)
Population: The pharmacokinetic (PK) parameter analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "n" signifies participants who were evaluable at the specified time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | ReFacto AF: Less Than 6 Years | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 18 | 19
(IU/dL)/(IU/kg)
  Day 1 (n= 17, 18) | 1.67 (0.361) | 1.97 (0.437)
  Day 15 (n= 18, 17) | 1.23 (0.650) | 1.91 (0.423)
  Day 50 (n= 17, 18) | 1.66 (0.626) | 1.96 (0.586)
  Month 6 (n= 2, 5) | 1.69 (0.210) | 2.17 (0.379)
  Month 18 (n= 4, 5) | 1.81 (0.405) | 1.80 (0.493)
  Final Visit (n= 17, 17) | 1.98 (1.454) | 1.89 (0.503)

3. Primary Outcome: Terminal Elimination Half Life of ReFacto AF (t1/2)
Description: T1/2 was the time for the plasma concentration of drug to decrease by one-half of its original concentration.
Time Frame: Pre-dose, 0.5, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose on Day 1
Population: PK parameter analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure. Data was not planned to be collected and analyzed for reporting arm "ReFacto AF: Less Than 6 Years", as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 14
hours | 9.12 (1.9429)

4. Primary Outcome: Clearance (CL)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose, 0.5, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour per kilogram
Arm/Group | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 14
milliliter per hour per kilogram | 4.406 (30)

5. Secondary Outcome: Mean Annualized Bleeding Rates (ABRs): All Participants
Description: ABR for each participant was calculated as the number of bleeds requiring administration of FVIII replacement product (taken from the Infusion Log Diary case report form), divided by the total therapy duration (in days), then multiplied by 365.25. ABR for the participants who reported following a primary or secondary prophylaxis, on-demand regimen or preventive regimen at baseline were reported.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: bleeds per year
Groups:
- ReFacto AF: All Participants: All participants (aged less than or equal to [<=] 12 years of age) were treated with IV injections of ReFacto AF at a dose and frequency prescribed by the investigator (minimum dose of 17 IU/kg up to maximum dose of 51 IU/kg) as per local standard of care in accordance with the SmPC.
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 36
bleeds per year
  On-demand regimen (n=14) | 27.51 (20.387)
  Preventive regimen (n=0) | NA (NA) — Data was not calculated and reported because none of the participants were reported at baseline as following a preventive regimen.
  Primary or secondary prophylaxis regimen (n=22) | 4.18 (3.849)

6. Secondary Outcome: Response to First On-Demand Treatment for New Bleeds: All Participants
Description: A 4-point scale of assessment of 'on-demand' treatment (administration of an unscheduled bolus infusion of Refacto-AF to stop bleeding) is defined as: 1. Excellent: Definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with no additional infusion administered. 2. Good: Definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with at least one additional infusion administered for complete resolution of the bleeding episode;or, Definite pain relief and/or improvement in signs of bleeding starting after 8 hours following infusion, with no additional infusion administered. 3. Moderate: Probable or slight improvement starting after 8 hours following the infusion, with at least one additional infusion administered for complete resolution of the bleeding episode. 4. No Response: No improvement at all between infusions or during the 24-hour interval following an infusion, or condition worsens.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure and received at least 1 dose of ReFacto AF for at least one bleeding episode.
Measure: Number; unit: responses
Units Other Than Participants: bleeds
Groups:
- ReFacto AF: All Participants: All participants (aged <=12 years of age) were treated with IV injections of ReFacto AF at a dose and frequency prescribed by the investigator (minimum dose of 17 IU/kg up to maximum dose of 51 IU/kg) as per local standard of care in accordance with the SmPC.
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 30
Number analyzed (bleeds) | 804
responses
  Excellent | 713 (20.387)
  Good | 73 (NA)
  Moderate | 16 (3.849)
  Data Not Recorded | 2

7. Secondary Outcome: Number of On-Demand ReFacto AF Infusions to Treat a New Bleed: All Participants
Description: The infusion log diary case report form (CRF) was used to determine the number of on-demand (administration of an unscheduled bolus infusion of Refacto-AF to stop bleeding) ReFacto AF infusions administered to treat a new bleed. This was calculated by adding the initial for a new bleed (on-demand) infusion to any subsequent (on-demand) infusions for the same "previously treated bleed" (same bleed with same start date/time).
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: infusions
Units Other Than Participants: bleeds
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 30
Number analyzed (bleeds) | 804
infusions | 1.1 (0.55)

8. Secondary Outcome: Number of Breakthrough Bleeds Within 48 Hours of a Prophylaxis Dose of ReFacto AF: All Participants
Description: The number of breakthrough bleeds within 48 hours following a prophylaxis dose of ReFacto AF was summarized. The infusion log diary CRF was used to determine the number of infusions administered to treat a new bleed counting only those infusions which were administered <=48 hours after an infusion marked as "prophylaxis" (which had no associated bleed).
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: breakthrough bleeds
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
breakthrough bleeds | 2.0 (1.15)

9. Secondary Outcome: Average Infusion Dose of ReFacto AF: All Participants
Description: The average infusion dose (by weight) for each participant was calculated as his total factor FVIII consumption (in IU) divided by weight (in kg) divided by the number of infusions administered in total study duration. Data was reported separately for participants classified at baseline as following non-prophylaxis regimen (for example: on-demand regimen, preventive, or not specified), and participants classified at baseline following a primary or secondary prophylaxis regimen.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "n" signifies participants who were evaluable for each specified baseline category.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
IU/kg
  With prophylaxis regimen at baseline (n= 22) | 37.0 (8.70)
  With non-prophylaxis regimen at baseline (n= 15) | 29.5 (7.61)

10. Secondary Outcome: Total Factor VIII Consumption: All Participants
Description: Total factor VIII consumption for each participant was calculated by sum of the total amount of ReFacto AF (in IU) infused for each ReFacto AF infusion (recorded in the infusion log diary CRF). Data was reported separately for participants classified at baseline as following non-prophylaxis regimen (for example: on-demand regimen, preventive, or not specified), and participants classified at baseline following a primary or secondary prophylaxis regimen.
Time Frame: Baseline up to Month 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
IU
  With Prophylaxis regimen at baseline (n= 22) | 97959.4 (48474.09)
  With non-prophylaxis regimen at baseline (n= 15) | 84051.7 (47362.60)

11. Secondary Outcome: Number of Less-Than-Expected-Therapeutic Effect (LETE) Bleeds in the On-Demand Setting: All Participants
Description: LETE in on-demand setting was based on response to treatment of a bleeding episode. LETE in the on-demand setting occurred if participant recorded 2 successive "no response" ratings after 2 successive ReFacto AF infusions. Both infusions were to be administered at an interval of 24 hours for treatment of same bleeding event in absence of confounding factor which included: known presence or subsequent identification of a FVIII inhibitor, known inadequate dose for type and/or severity of bleed in opinion of investigator, delay of greater than 4 hours between onset of bleed to infusion, delay of greater than 24 hours before administration of a follow-up infusion, known compromised ReFacto AF, faulty administration of ReFacto AF, participant had an underlying, predisposing condition responsible for bleed in opinion of investigator (e.g., kidney stones or use of medications known to impair platelet function, such as aspirin or NSAIDs),or ongoing trauma responsible for continued bleeding.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure and received treatment for at least one bleed.
Measure: Number; unit: LETE bleeds
Units Other Than Participants: bleeding episodes
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 30
Number analyzed (bleeding episodes) | 804
LETE bleeds | 0

12. Secondary Outcome: Number of Less-Than-Expected-Therapeutic Effect (LETE) Bleeds in the Prophylaxis Setting: All Participants
Description: LETE in the prophylaxis setting occurred if there was a spontaneous bleed within 48 hours (<=48 hours) after a regularly scheduled prophylactic dose of ReFacto AF (which was not used to treat a bleed) in the absence of confounding factors. Therefore, LETE in the prophylaxis setting is the occurrence of a bleed. Confounding factors include: Known presence or subsequent identification of a FVIII inhibitor, known inadequate prophylactic dose, known lack of adherence to the prescribed prophylaxis regimen, bleed occurs in a target joint identified at the start of the study, known compromised ReFacto AF, faulty administration of ReFacto AF, an underlying, predisposing condition responsible for the bleed in the opinion of the investigator (e.g., kidney stones or use of medications known to impair platelet function, such as aspirin or NSAIDs) or traumatic injury responsible for bleeding.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Participants who received at least 1 prophylaxis dose of ReFacto AF were reported.
Measure: Number; unit: LETE bleeds
Units Other Than Participants: prophylaxis infusions
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
Number analyzed (prophylaxis infusions) | 2457
LETE bleeds | 2

13. Secondary Outcome: Number of Occurrences of Less-Than-Expected-Therapeutic Effect (LETE) in the Low Recovery Setting: All Participants
Description: LETE in the low recovery setting was defined as lower than expected recovery of FVIII (in the opinion of investigator), following the infusion of ReFacto AF in the absence of confounding factors for the low recovery. The only confounding factors for low recovery are as follows: known presence or subsequent identification of a FVIII inhibitor, known compromised ReFacto AF, faulty administration of ReFacto AF, including inadequate dosing.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF.
Measure: Number; unit: LETE bleeds
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
LETE bleeds | 9

14. Secondary Outcome: Number of Participants Requiring Escalated Dose of Prescribed Regimen During the Treatment Period: All Participants
Description: Participants who met the dose escalation criteria were prescribed a higher dose and/or more frequent doses as per the investigator's discretion.
Time Frame: Baseline up to Month 24
Population: Efficacy analysis population included all enrolled participants who received at least 1 dose of ReFacto AF. Participants who used a prophylaxis regimen were analyzed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
participants | 5

15. Secondary Outcome: Plasma Concentration of Factor VIII at 0.5 Hour Post-dose (C0.5)
Time Frame: 0.5 hour post-dose on Day 1
Population: The PK parameter analysis population included all enrolled participants who received at least 1 dose of ReFacto AF.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | ReFacto AF: Less Than 6 Years | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 18 | 19
IU/mL | 0.752 (18) | 0.903 (45)

16. Secondary Outcome: Area Under the Plasma Time Curve From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: AUCinf is the area under the plasma concentration-time profile from time 0 extrapolated to infinite time. It was calculated as International units*hour per milliliter (IU*hr/mL).
Time Frame: Pre-dose, 0.5, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 14
IU*hr/mL | 9.89 (41)

17. Secondary Outcome: Area Under the Plasma Time Curve From Time Zero to Time of Last Measurable Concentration (AUClast)
Description: AUClast is the area under the plasma versus time curve from time zero to time of last measurable concentration (AUClast)
Time Frame: Pre-dose, 0.5, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 14
IU*hr/mL | 9.49 (41)

18. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug was uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) was the apparent volume of distribution at steady-state.
Time Frame: Pre-dose, 0.5, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 14
mL/kg | 56.42 (15)

19. Secondary Outcome: Mean Residence Time (MRT) of ReFacto AF
Description: MRT was calculated as AUMCinf / AUCinf-TI/2, where AUMCinf is the area under the first moment curve from time zero to infinity and TI was the duration of infusion.
Time Frame: Pre-dose, 0.5, 1, 3, 6, 9, 24, 28, 32, 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | ReFacto AF: 6 to Less Than 12 Years
Number analyzed (Participants) | 14
hour | 13.91 [8.51 to 18.3]

20. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): All Participants
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 30 days after last study visit (Month 25)
Population: Safety analysis population included all enrolled participants who received at least 1 dose of ReFacto AF.
Measure: Number; unit: participants
Arm/Group | ReFacto AF: All Participants
Number analyzed (Participants) | 37
participants
  AEs | 28
  SAEs | 6

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last study visit (Month 25)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and nonserious in another participant, or one participant may have experienced both serious and nonserious event during study. Adverse events data was planned to be reported for overall population.
Arm/Group | ReFacto AF: All Participants
Serious Adverse Events (participants affected / at risk) | 6/37
Other Adverse Events (participants affected / at risk) | 28/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReFacto AF: All Participants (N=37)
Factor VIII inhibition (Blood and lymphatic system disorders) | 4
Laryngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Scrotal disorder (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReFacto AF: All Participants (N=37)
Nasopharyngitis (Infections and infestations) | 12
Influenza (Infections and infestations) | 3
Adenoiditis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Otitis media acute (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Cestode infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pyoderma streptococcal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 4
Head injury (Injury, poisoning and procedural complications) | 4
Joint injury (Injury, poisoning and procedural complications) | 3
Limb injury (Injury, poisoning and procedural complications) | 2
Tooth fracture (Injury, poisoning and procedural complications) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Lip haemorrhage (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Oral cavity fistula (Gastrointestinal disorders) | 1
Tooth pulp haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 3
Hypotension (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Underweight (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Solar urticaria (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.